CLINICAL TRIAL: NCT01618136
Title: An Open-Label, Multicenter, Phase 1/2 Study of Poly(ADP-Ribose) Polymerase (PARP) Inhibitor E7449 as Single Agent in Subjects With Advanced Solid Tumors or With B-cell Malignancies and in Combination With Temozolomide (TMZ) or With Carboplatin and Paclitaxel in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7449-E044-101
Record Dates: First submitted 2012-05-14; First posted 2012-06-13 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2016-10

CONDITIONS: Malignant Solid Tumour; Ovarian Cancer; Triple Negative Breast Cancer; Advanced Melanoma; B-cell Malignancy, Low-grade
Keywords: PARP inhibitors; Malignant Solid Tumour; ovarian cancer; triple negative breast cancer; advanced melanoma
MeSH Terms: conditions — Ovarian Neoplasms; Triple Negative Breast Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — stenoparib; Temozolomide; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- E7449 (Experimental)
  Interventions: Drug: E7449 alone
- E7449 plus TMZ (Active Comparator)
  Interventions: Drug: E7449 plus TMZ
- E7449 plus carboplatin and paclitaxel (Active Comparator)
  Interventions: Drug: E7449 plus carboplatin and paclitaxel

INTERVENTIONS:
Drug: E7449 alone — Will be administered as single agent orally, once daily (QD) continuously in 28-day cycles to determine the MTD. In these subjects, a food-effect component will be conducted under fed/fasted conditions to determine the effect of food on the bioavailability of E7449 administered orally QD.
  Arms: E7449
Drug: E7449 plus TMZ — Dose escalation,will be administered orally, once daily for 7 consecutive days along with 150 mg/m2/d TMZ administered orally, once daily for 5 consecutive days in 28-day cycles to determine the MTD of E7449 in combination with TMZ.
  Arms: E7449 plus TMZ
Drug: E7449 plus carboplatin and paclitaxel — Dose escalation, E7449 will be administered orally, once daily continuously in 21-day cycles along with carboplatin and paclitaxel, which will be administered via i.v. infusion on Day 1 of the cycle only, to determine the MTD of E7449 in combination with carboplatin and paclitaxel.
  Arms: E7449 plus carboplatin and paclitaxel

SUMMARY:
Overall Design: This is a multicenter, open-label, Phase 1/2 study which will be conducted in three arms (as described below). Each arm will be conducted in two parts: a Phase 1 part which will include dose escalation and a Phase 2 part which will include four cohorts in specific disease indications. Phase 1 will also include a food effect study of E7449 as a single agent. Once the MTD in the Phase 1 single agent arm and the Phase 1 combination arms of this study has been achieved, the sponsor will submit the relevant safety information and recommended Phase 2 dose to the IRB/Health Authorities. Arm 1: E7449 will be administered as a single agent. Arm 2: E7449 will be administered in combination with TMZ. Arm 3: E7449 will be administered in combination with carboplatin and paclitaxel

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Subjects with measurable or non-measurable disease following the Response Evaluation Criteria in Solid Tumors (RECIST 1.1, Appendix 1) for Phase 1 part of the study. (Only subjects with measurable disease are allowed to enter at the MTD during the expanded cohort of Phase 1)
2. Histologically and/or cytologically confirmed advanced or metastatic solid tumor or Bcell malignancies which have progressed after treatment with approved therapies or for which there are no standard therapies available (Phase 1).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Appendix 2).
4. Life expectancy greater than or equal to 3 months after starting E7449.
5. Subjects with known brain metastases will be eligible under the following conditions (see Exclusion Criterion #2):

   * has undergone complete surgical excision and are more than 1 month post surgery with no radiographic evidence of brain disease recurrence Or
   * has undergone stereotactic radio surgery (gamma knife procedure) and are more than 1 month post procedure and with no radiographic evidence of brain disease progression And
   * is asymptomatic And
   * discontinued corticosteroid treatment at least 30 days prior to C1D1.
6. Adequate renal function defined as Serum Creatinine less than 1.5 x ULN, or use SI units or calculated creatinine clearance greater than or equal to 50 mL/min per the Cockroft-Gault formula (Appendix 3).
7. Adequate bone marrow function:

   * Absolute neutrophil count (ANC) greater than or equal to1500/mm3 (greater than or equal to 1.5 x 10^3/mL);
   * Platelets greater than or equal to 100,000/mm3 (greater than or equal to 100 x 10^9/L);
   * Hemoglobin greater than or equal to 10.0 g/dL.
8. Adequate liver function:

   * Bilirubin less than or equal to 1.5 x the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome;
   * Alkaline phosphatase (in the absence of bone disease), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 x ULN (less than or equal to 5 x ULN if subject has liver metastasis).
9. Left ventricular ejection fraction (LVEF) greater than 50% on echocardiography or multiple-gated acquisition (MUGA) scanning
10. Males or females age greater than or equal to 18 years at the time of informed consent.
11. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [beta-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of beta-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug. All females will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrheic, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing). Females of childbearing potential must not have had unprotected sexual intercourse within 30 days prior to study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the subject must agree to use a double-barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
12. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partner must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation).
13. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

    For the Phase 2 Cohort 1 (Platinum-sensitive recurrent high-grade serous ovarian cancer) only:
14. Histologically confirmed platinum-sensitive recurrent high grade serous ovarian cancer locally advanced or metastatic with disease progression after standard treatments. (Exclude platinum refractory/resistant defined as progression on platinum or relapse within six months of prior platinum.
15. At least one lesion of greater than or equal to 1.0 cm in the longest diameter for a non-lymph node or greater than or equal to 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI) or photography. If there is only one target lesion, it should have a longest diameter of greater than or equal to 1.5 cm (for a non-lymph node) or greater than or equal to 1.5 cm in the short-axis diameter (for a lymph node).

    For the Phase 2 Cohort 2 (B-cell malignancies) Only:
16. Subjects with one of the following relapsed and/or refractory B-cell malignancies with disease progression following up to three prior systemic treatment regimens:

    * Mantle cell, Marginal zone, Follicular, Diffuse large B-cell, B-cell chronic lymphocytic leukemia (B-CLL).
    * ATM-deficient.

    For the Phase 2 Cohort 3 (Melanoma) only:
17. Histopathologically confirmed advanced melanoma (except melanoma of intraocular origin) with disease progression following up to two systemic treatment regimens
18. At least one lesion of greater than or equal to 1.0 cm in the longest diameter for a non-lymph node or greater than or equal to 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI) or photography. If there is only one target lesion, it should have a longest diameter of greater than or equal to 1.5 cm (for a non-lymph node) or greater than or equal to 1.5 cm in the short-axis diameter (for a lymph node).
19. No previous treatment with dacarbazine (DTIC) or TMZ containing regimens

    For the Phase 2 Cohort 4 (mTNBC) only:
20. Histologically confirmed metastatic triple-negative breast cancer. Estrogen receptor (ER)-negative, Progesterone Receptor (PR)-negative, Human Epidermal Growth Factor 2 (HER2)-negative (mTNBC) with disease progression after one standard treatment.
21. At least one lesion of greater than or equal to 1.0 cm in the longest diameter for a non-lymph node or greater than or equal to 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI) or photography. If there is only one target lesion, it should have a longest diameter of greater than or equal to 1.5 cm (for a non-lymph node) or greater than or equal to 1.5 cm in the short-axis diameter (for a lymph node).
22. No previous treatment with carboplatin and/or paclitaxel.

Exclusion Criteria:

All subjects

1. Prior exposure to E7449.
2. Leptomeningeal metastases or brain metastases (except as for Inclusion Criterion #5).
3. Prior treatment with a PARP inhibitor (Phase 2 only).
4. Subjects taking medications which are either strong CYP inhibitors or inducers.
5. Subjects with active malignancies other than advanced ovarian cancer (Cohort 1 only), ATM-deficient B-cell malignancies (Cohort 2 only), advanced melanoma (Cohort 3 only), and mTNBC (Cohort 4 only), will be excluded from Phase 2.
6. Subjects who have received any anticancer treatment within 4 weeks or any investigational agent within 30 days prior to the first dose of study drug or who have not recovered from any acute toxicity greater than Grade 0 or 1 related to previous anticancer treatment.
7. Major surgery within 4 weeks prior to the first dose of study drug.
8. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of E7449.
9. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment.
10. Prolongation of QTc interval to greater than 480 msec when electrolytes balance is normal.
11. Active infection requiring systemic therapy.
12. Known hypersensitivity to any component of E7449
13. Achlorhydria or use of antacids, proton-pump inhibitors, or other drugs known to raise gastric pH within 2 weeks prior to study drug administration.
14. Other relevant disease or adverse clinical conditions such as:

    History of significant neurological (no neuropathy greater than Grade 2) or psychiatric disorders.
    * Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).
    * Significant non-neoplastic renal disease.
    * Immunocompromised patients, including patients known to be infected with human immunodeficiency virus (HIV).
    * Uncontrolled endocrine diseases (e.g., diabetes mellitus, hypothyroidism or hyperthyroidism, adrenal disorder) i.e., requiring relevant changes in medication within the last month or hospital admission within the last three months.
    * Tumor bleeding
15. Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study
16. Females who are pregnant or breastfeeding.

    For Phase 1 Arm 2 and Phase 2 Arm 2 (E7449 in combination with TMZ) only:
17. Known intolerance or known hypersensitivity to any of the study drugs or any of the Excipients (E7449 and/or TMZ) For Phase 1 Arm 3 and Phase 2 Arm 3 (E7449 in combination with carboplatin and paclitaxel) only:
18. Known intolerance or known hypersensitivity reactions to E7449, carboplatin or other platinum containing compounds, paclitaxel, macrogolglycerol ricinoleate (poloxyl castor oil) or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Phase 1 To determine the maximum tolerated dose of E7449 as a single agent | Baseline to 24 months.
Phase 1 To determine the maximum tolerated dose of E7449 and in combination with TMZ | Baseline to 24 months.
Phase 1 To determine the maximum tolerated dose of E7449 and in combination with carboplatin and paclitaxel | Baseline to 24 months.

SECONDARY OUTCOMES:
Phase 2 to assess the objective response rate of E7449 as a single agent in subjects with platinum sensitive recurrent high-grade serious ovarian cancer and subjects with relapsed and/or refractory ATM- deficient B-cell malignancies | Baseline to 20 months.
Phase 2 to assess the objective response rate of E7447 in combination with TMZ in subjects with advanced melanoma | Baseline to 20 months.
Phase 2 to assess the objective response rate of E7449 in combination with carboplatin and paclitaxel in subjects with metastatic triple negative breast cancer | Baseline to 20 months.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - King's College London Guy's Hospital Campus, London
  - Newcastle Upon Tyne NHS Foundation Trust, Newcastle Upon Tyne and Wear

REFERENCES:
- [Derived] Plummer R, Dua D, Cresti N, Drew Y, Stephens P, Foegh M, Knudsen S, Sachdev P, Mistry BM, Dixit V, McGonigle S, Hall N, Matijevic M, McGrath S, Sarker D. First-in-human study of the PARP/tankyrase inhibitor E7449 in patients with advanced solid tumours and evaluation of a novel drug-response predictor. Br J Cancer. 2020 Aug;123(4):525-533. doi: 10.1038/s41416-020-0916-5. Epub 2020 Jun 11. PMID 32523090